CLINICAL TRIAL: NCT00751309
Title: Lung Allograft Rejection Gene Expression Observational (LARGO) Study
Acronym: LARGO
Status: Terminated | Type: Observational
Why Stopped: Restructuring and refocus of company.
Sponsor: XDx (Industry)
Responsible Party: Kenneth C. Fang, MD, XDx, Inc.
Other Study IDs: LARGO
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Graft Rejection; Lung Disease
Keywords: allograft; rejection; biopsy; gene; expression; pulmonary; lung; transplant
MeSH Terms: conditions — Lung Diseases; Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Lung and heart-lung transplanted subjects.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Post-transplantation observational study

SUMMARY:
The objective of the LARGO Study protocol is to collect peripheral blood samples, select associated lung biopsy pathology slides, and clinical data from lung transplant recipients to perform molecular analyses in association with the study endpoints. The primary objective is to use gene expression profiling of peripheral blood mononuclear cells to differentiate between the absence and presence of acute cellular rejection. The secondary objectives are to use other genomic and proteomic technologies to analyze RNA and protein in blood samples in relation to related clinical conditions. The overall goal is to apply novel molecular insights in the development of non-invasive molecular diagnostic tests for lung transplantation.

DETAILED DESCRIPTION:
LARGO is a prospective, multi-center, international observational study with participating centers in the United States, Canada and Europe. The target enrollment for study completion is 2,100 subjects.

At each study visit, blood specimens are collected from subjects, processed and stored in the sample archive, with corresponding patient information entered into the clinical database. The analysis plan for each study objective includes a defined sample selection protocol that stipulates the inclusion and exclusion criteria for both patients and samples, and also the required number of blood specimens for the molecular analyses to achieve statistical significance.

The diagnosis and treatment of acute cellular rejection remains a clinical management priority that is currently based on transbronchial biopsy. Gene expression profiling is a technology based on molecular biology that measures changes in the RNA levels of different genes expressed by circulating mononuclear cells in the peripheral blood. A key goal of the project is to use gene expression profiling to differentiate between the absence and presence of lung allograft acute cellular rejection, with the aim of using this novel information to develop a non-invasive diagnostic testing alternative.

ELIGIBILITY:
Inclusion Criteria:

* Lung and heart-lung transplant recipients who consent to participate and have transbronchial biopsy at the enrolling center during the study period

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Lung and heart-lung transplant recipients who will undergo transbronchial biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 2044 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Rejection episodes of at least moderate histologic grade which resulted in treatment of the patient with additional corticosteroids, anti-T cell antibodies, or total lymphoid irradiation. | Scheduled clinic visit
Obliterative Bronchiolitis diagnosed pathologically by biopsy or by a progressive decline in pulmonary function tests consistent with a diagnosis of Bronchiolitis Obliterans Syndrome (BOS). | Scheduled clinic visit
Allograft function as determined via pulmonary function tests. | Scheduled clinic visit
The absence of histologic rejection and normal or unchanged allograft function. | Scheduled clinic visit
Documented CMV infection by culture, histology, or PCR, and at least one clinical sign or symptom of infection. | Scheduled clinic visit
Infections other than CMV, e.g. bacterial, other viral, and fungal infections. | Scheduled clinic visit

SECONDARY OUTCOMES:
Rejection of mild to moderate histologic severity prompting augmentation of the patient's chronic immunosuppressive regimen. | Scheduled clinic visit
Allograft dysfunction during the study period. | Scheduled clinic visit
Rejection of mild to moderate severity with allograft dysfunction prompting plasmapheresis or a diagnosis of "humoral" rejection. | Scheduled clinic visit
Lymphoproliferative disorder (aka post-transplant lymphoma). | Scheduled clinic visit
Graft Failure or Retransplantation. | Scheduled clinic visit
All cause mortality. | Scheduled clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C. Fang, MD, Study Director — XDx, Inc.
Locations (20):
- United States (15):
  - UCLA Division of Pulmonary and Critical Care, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Transplant Center, Jacksonville, Florida
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University College of Physicians and Surgeons, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - University Hospital and Clinics, Madison, Wisconsin
- Medizinische Universität Wien, Vienna, Austria
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Medizinische Hochschule Hannover, Hanover, Germany
- Freeman Hospital, High Heaton, Newcastle upon Tyne, United Kingdom

REFERENCES:
- See also: Information on molecular expression testing — http://www.xdx.com/allomap
- See also: Sponsor's website — http://www.xdx.com